CLINICAL TRIAL: NCT05585398
Title: A Phase 1 Single-center Study to Evaluate the Distribution of NT 201 Administered as Intradermal Injections, Comparing Different Doses, Concentrations, and Delivery Methods
Brief Title: A Study to Evaluate the Distribution of Botulinum Neurotoxin Type A Administered as Intradermal Injections, Comparing Different Doses, Concentrations, and Delivery Methods
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merz Pharmaceuticals GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M602011074; 2021-005901-29 (EudraCT Number)
Record Dates: First submitted 2022-10-14; First posted 2022-10-18 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: N/A, as no Specific Medical Condition Will be Treated
MeSH Terms: interventions — incobotulinumtoxinA; Botulinum Toxins, Type A

STUDY DESIGN:
Intervention Model Description: Intra-individual comparison
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- LMRC (left with micro-/right with conv- needle) (Experimental)
  Interventions: Drug: IncobotulinumtoxinA
- RMLC (right with micro-/left with conv- needle) (Experimental)
  Interventions: Drug: IncobotulinumtoxinA
- LCRM (left with conv-/ right with micro-needles) (Experimental)
  Interventions: Drug: IncobotulinumtoxinA
- RCLM (right with conv-/left with micro-needles) (Experimental)
  Interventions: Drug: IncobotulinumtoxinA

INTERVENTIONS:
Drug: IncobotulinumtoxinA — Intradermal injections using different delivery methods (conventional needle and microneedles)
  Other Names: Xeomin; Botulinum toxin type A (150 kiloDalton), free from complexing proteins

SUMMARY:
The purpose of this study is to evaluate the distribution of IncobotulinumtoxinA (Xeomin) in healthy subjects at different volumes, concentrations and doses when administered intradermally and subcutaneously using different delivery methods (conventional needle and microneedles).

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subject aged 18 to 45 years with body mass index (BMI) 19.0 to 27.0 kg/m².
* Subject with the distance not less than 45 cm between the spinous process of the 7th cervical vertebra (C7) and the 4th lumbar vertebra (L4).
* Healthy skin at test area (forehead and back).
* Fitzpatrick skin type I to IV.
* Displaying uniform sweating activity (i.e., symmetrical sweating pattern with enough sweat and without anhidrotic regions) on the forehead area as assessed with Minor's starch iodine test under standardized sweating conditions.

Exclusion Criteria:

* Any chronic pain conditions or presence of acute pain of any origin and intensity.
* Dermal treatment of the forehead (e.g., light resurfacing, dermabrasions) within the last 12 months before Screening, during the screening period, and/or at Baseline.
* Any type of filler in the treatment area on the facial region within the last 12 months before Screening, during the screening period, and/or atBaseline; regardless of time for any type of implant and/or surgery in the treatment area on facial region.
* Any type of surgery in the treatment area of the back within the last 12 months before Screening, during the screening period, and/or at Baseline.
* Treatment with anticholinergics within the last 14 days before Screening, during the screening period, and/or at Baseline.
* Treatment with analgesics (e.g., non steroidal anti inflammatory drugs, except acetylsalicylic acid, ibuprofen, and paracetamol) within the last 10 days before Screening, during the screening period, and/or prior to pain assessment at Baseline.
* Treatment with paracetamol, ibuprofen, or acetylsalicylic acid within three days prior to pain assessment at Baseline.
* Subjects with excessive sweating or previously diagnosed with hyperhidrosis.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-10-19 (Actual); Primary Completion 2023-02-24 (Actual); Study Completion 2023-04-13 (Actual)

PRIMARY OUTCOMES:
Area of anhidrosis on contralateral points of the forehead four weeks after intradermal injections of NT 201 with fixed dose and volume, using different delivery methods | Week 4

SECONDARY OUTCOMES:
Injection pain intensity as assessed by a 0-10 numeric pain rating scale directly after the intradermal injection of NT 201 applied via different delivery methods in the forehead | Week 4

CONTACTS AND LOCATIONS:
Overall Officials: Merz Medical Expert, Study Director — Merz Therapeutics GmbH
Locations (1):
- Merz Investigational Site #0490385, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No